CLINICAL TRIAL: NCT00028522
Title: Phase I Study Of R(+)XK469 In Patients With Advanced Neuroblastoma
Brief Title: R(+)XK469 in Treating Patients With Advanced Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00013; NCI-2009-00013 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-11108B; CDR0000739128; NCI-4570; 11108B (Other: University of Chicago Comprehensive Cancer Center); 4570 (Other: CTEP); U01CA069852 (NIH)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Disseminated Neuroblastoma; Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — XK 469

ARMS (1):
- Treatment (chemotherapy) (Experimental): SCHEDULE A: Patients receive R(+)XK469 IV over 30 minutes on days 1, 3, and 5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of R(+)XK469 until the recommended phase II dose or MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued and treated at the recommended phase II dose (for a maximum of 20 patients treated at that dose).
  SCHEDULE B: Once the recommended phase II dose is determined on schedule A, additional patients are accrued and receive escalating doses of R(+)XK469 IV over 30-60 minutes on day 1, beginning at a reduced dose. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Dose escalation continues as in Schedule A.
  Interventions: Drug: R(+)XK469

INTERVENTIONS:
Drug: R(+)XK469 — Given IV
  Other Names: XK469

SUMMARY:
This phase I trial is studying the side effects and best dose of R(+)XK469 in treating patients with advanced neuroblastoma. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose, recommended phase II dose, and dose-limiting toxicity of R(+)XK469 in two different dosing schedules in patients with advanced neuroblastoma.

II. Determine the safety of this drug in these patients. III. Determine the tolerance to this drug in these patients. IV. Determine the pharmacokinetics and pharmacodynamics of this drug and its metabolites in these patients.

V. Determine, preliminarily, any antineoplastic activity of this drug in these patients.

OUTLINE: This is a dose-escalation study.

SCHEDULE A: Patients receive R(+)XK469 intravenously (IV) over 30 minutes on days 1, 3, and 5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of R(+)XK469 until the recommended phase II dose or maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued and treated at the recommended phase II dose (for a maximum of 20 patients treated at that dose).

SCHEDULE B: Once the recommended phase II dose is determined on schedule A, additional patients are accrued and receive escalating doses of R(+)XK469 IV over 30-60 minutes on day 1, beginning at a reduced dose. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Dose escalation continues as in Schedule A.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-risk neuroblastoma that has relapsed or is refractory to standard therapy
* No active brain metastases

  * Previously treated brain metastases allowed if there is no requirement for corticosteroids or anticonvulsants
* Performance status - Karnofsky performance status 70-100% or Lansky score ≥ 70 for your pediatric patients
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal (unless due to documented Gilbert's syndrome)
* Creatinine less than 1.5 times upper limit of normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent uncontrolled illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No prior allergic reaction to compounds of similar chemical or biological composition to study drug (e.g., flurbiprofen or ibuprofen)
* No HIV-positive patients
* No concurrent biologic agents
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* No other concurrent chemotherapy
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy
* See Disease Characteristics
* Recovered from all prior therapy
* No other concurrent investigational agents
* No concurrent commercial agents or therapies directed at malignancy
* No concurrent combination anti-retroviral therapy for HIV-positive patients

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2001-12; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of XK469 in pediatric patients with advanced neuroblastoma | Day 29 of course 1
  Defined as the highest dose studied for which the incidence of dose-limiting toxicity (DLT) was less than 33%.
DLT | Day 29 of course 1
  Defined as the occurrence of any of the following: 1) grade 3 or higher nonhematologic toxicity except fatigue, alopecia, nausea, vomiting, 2) grade 4 thrombocytopenia or anemia, 3) any fever accompanied by granulocyte count < 1000/mm^3 (grade 3 or 4 neutropenia), 4) failure to recover absolute neutrophil count 1500/μL
Recommended phase II dose | Day 29 of course 1
  Generally defined as the MTD. For both schedules A and B and the pediatric dosing schedule, once the recommended phase II dose has been tentatively defined, a total of 12 evaluable patients will be studied to ensure the feasibility of this dose for phase II trials. If interindividual pharmacokinetic variability is high, additional patients will be enrolled (maximum of 20 at the phase II dose) to permit adequate pharmacological characterization of XK469 and the relationship of interindividual pharmacokinetic variability to toxicity.

SECONDARY OUTCOMES:
Metabolism of XK469 in pediatric patients | Days 1-3 of course 1
  Performed by high-performance liquid chromatography (HPLC). Plasma metabolic ratios between metabolite and XK469 concentrations will be used as an index of metabolic activity and phenotype for each patient. The modality of the frequency distribution of metabolic ratios will be also described.
Pharmacokinetics of XK469 in pediatric patients | Days 1-3 of course 1
  The maximum number of samples for pharmacokinetic studies will not exceed 20. Analyzed by non compartmental method using the WinNonlin software. Parameters include the elimination rate constant, the area under the concentration vs. time curve (AUC), terminal half-life, total (nonrenal + renal) clearance, and volume of distribution at steady state. Mean, standard deviation, and coefficient of variation will be determined for each parameter.
Pharmacodynamics of XK469 in pediatric patients | Continuously over the course of study treatment
  Performed by correlating area under the curve (AUC) (and other parameters) of R(+)XK469 and metabolites with observed toxicities. Specifically, we will compare the AUC in those patients who experience grade >= 2 toxicity to those who experience grade < 2 toxicity using a Wilcoxon, nonparametric rank-sum test.
Antineoplastic activity of XK469 for neuroblastoma | Every 2 courses
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Cohn, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States